CLINICAL TRIAL: NCT02801292
Title: Ketamine as an Adjuvant Therapy for Acute Vaso Occlusive Crisis in Pediatric Patients With Sickle Cell Disease, a Pilot Study
Brief Title: Ketamine as an Adjuvant Therapy for Acute Vaso Occlusive Crisis in Pediatric Patients With Sickle Cell Disease
Acronym: KSickle
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 917282
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- administering of ketamine (Other): adjuvant to standard of care
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Single bolus of Ketamine .25 milligrams per kilogram of weight.
  Other Names: ketamine hydrochloride

SUMMARY:
The primary objective of the proposed study is to determine the potential role of Ketamine as an analgesic agent in pediatric sickle cell disease patients with refractory symptoms in acute (VOC).

DETAILED DESCRIPTION:
The primary objective of the proposed study is to determine the potential role of Ketamine as an analgesic agent in pediatric sickle cell disease patients with refractory symptoms in acute (VOC). Our study design is as follows: Prospective observational study of 20 pediatric sickle cell disease patients with refractory pain to conventional analgesic regimens seen in the pediatric emergency medicine department. Consenting patients with refractory pain meeting inclusion criteria will be given a single intravenous bolus of Ketamine at a set dosage of 0.25 milligrams per kilogram of weight. Participants' perception of pain will then be recorded using standard pain scoring scales (FLACC score). Physiologic criteria such as heart rate, blood pressure, blood oxygen saturation, total analgesic pharmacologic requirements for adequate analgesia during hospitalization, and duration of hospitalization will be measured. Observational study group will continue to get standard of care outside of single bolus of Ketamine. 48 hour follow up after hospital discharge will be obtained to assess degree of pain control and general clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (> 3 yrs and <18yrs) with a previous diagnosis of sickle cell disease (including Hgb S Beta Thalassemia +, Hgb S Alpha Thalassemia, Hgb S HPFH) ) seen in the pediatric emergency room setting for acute vaso-occlusive pain crisis.

Exclusion Criteria:

* Patients not to have sequelae indicative of complicated disease outside of acute VOC:

  1. Acute chest syndrome (new pulmonary infiltrate and hypoxemia)
  2. Aplastic Episode
  3. Evidence of infection
  4. Pregnancy or CHF
  5. Fever (> 38.4)
  6. Cholangitis or cholecystitis
  7. Hypoxia (SaO2 <90% on RA), or O2 saturation decrease of more than 5% from patient's baseline
  8. Unstable Vital Signs
  9. Patients who have received intravenous pain medicine within 24 hours of visit to the emergency department.
  10. History of allergic reaction or serious reaction to Ketamine.
  11. History of significant psychiatric illness
  12. Patients with no refractory pain after receiving conventional analgesia regimen per protocol.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
pain score | 1 hour
  reduction in refractory pain

CONTACTS AND LOCATIONS:
Overall Officials: George Hsu, MD, Principal Investigator — Augusta University

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Background] Platt OS, Thorington BD, Brambilla DJ, Milner PF, Rosse WF, Vichinsky E, Kinney TR. Pain in sickle cell disease. Rates and risk factors. N Engl J Med. 1991 Jul 4;325(1):11-6. doi: 10.1056/NEJM199107043250103. PMID 1710777
- [Background] Koppert W, Sittl R, Scheuber K, Alsheimer M, Schmelz M, Schuttler J. Differential modulation of remifentanil-induced analgesia and postinfusion hyperalgesia by S-ketamine and clonidine in humans. Anesthesiology. 2003 Jul;99(1):152-9. doi: 10.1097/00000542-200307000-00025. PMID 12826855
- [Background] Mao J, Price DD, Mayer DJ. Mechanisms of hyperalgesia and morphine tolerance: a current view of their possible interactions. Pain. 1995 Sep;62(3):259-274. doi: 10.1016/0304-3959(95)00073-2. PMID 8657426
- [Background] Bergman SA. Ketamine: review of its pharmacology and its use in pediatric anesthesia. Anesth Prog. 1999 Winter;46(1):10-20. PMID 10551055